CLINICAL TRIAL: NCT00847327
Title: Parenting and Control Among Young Children With Type 1 Diabetes
Brief Title: Parental Management of Young Children's Diabetes
Acronym: YCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Children's National Research Institute (Other); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DK80102; R01DK080102 (NIH)
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Parenting; Young Children
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parental Support (Experimental)
  Interventions: Behavioral: Parental Support
- Diabetes Education (Active Comparator)
  Interventions: Behavioral: Diabetes Education

INTERVENTIONS:
Behavioral: Parental Support — The intervention utilizes cognitive behavioral strategies. Session 1 uses relaxation and cognitive reframing and explores parents' responses to the challenges of parenting a child with diabetes. Session 2 focuses on the emotional impact of having a child with diabetes and utilizes problem solving techniques. Session 3 focuses on child behavior and strategies for effective parenting. To facilitate support and community, Session 4 is a group session via conference call to discuss issues related to social support. Session 5 focuses on the impact diabetes has on the family and parents are taught cognitive reframing to help with managing diabetes. Parents are invited to participate in an Internet bulletin board moderated by trial personnel.
  Other Names: Cognitive Behavioral Strategies; Parent Support
  Arms: Parental Support
Behavioral: Diabetes Education — The education comparison group also participates in 5 sessions across 9 weeks. This group provides educational and resource support that is specific to managing diabetes in young children. Education topics include blood glucose monitoring, nutrition, and physical activity. Print materials are provided to participants and intervention sessions focus on talking points raised in these reading materials.
  Other Names: Diabetes Management; Nutrition; Exercise
  Arms: Diabetes Education

SUMMARY:
Type 1 diabetes is a lifelong metabolic disorder that affects 1 out of every 400-600 American children each year, with many children being diagnosed at younger and younger ages.

To achieve proper diabetes control, it is necessary to conform or adhere one's behavior to a physician-prescribed diabetes self-care regimen. As such, parents of children with Type 1 diabetes must be highly involved in managing their child's disease on a daily basis, especially parents of affected children who are very young and more highly dependent upon parental caretaking.

As children diagnosed with Type 1 diabetes at a very young age may be at an increased risk for the development of long-term behavioral and medical complications, more research is needed to understand and treat the leading contributors to diabetes-related parental distress and medical outcomes among this growing subgroup.

Recent findings indicate that responsibility for diabetes management falls heavily on mothers. The majority of families do not receive outside child care assistance and report feeling overwhelmed. Parents report high levels of pediatric parenting stress difficulty, as well as moderate symptoms of anxiety. The current study aims to expand such preliminary findings and specifically examine the effects of a newly-developed parenting support program for parents of young children with Type 1 diabetes. The utility of the intervention will be evaluated. It is hypothesized that parents completing the parent support program will report lower levels of psychosocial distress and improved quality of life. It is hypothesized that the children of participating parents will also demonstrate improved quality of life and metabolic control.

DETAILED DESCRIPTION:
Type 1 diabetes is a lifelong metabolic disorder that affects 1 out of every 400-600 American children each year, with many children being diagnosed at younger and younger ages. If Type 1 diabetes is not properly controlled, it can lead to a host of devastating disease-related complications later in life. Therefore, achieving proper diabetes control during childhood is an important public health issue.

To achieve proper diabetes control, it is necessary to conform or adhere one's behavior to a physician-prescribed diabetes self-care regimen consisting of multiple insulin administrations and blood glucose (BG) checks daily, as well as pay careful attention to diet and exercise. As such, parents of children with Type 1 diabetes must be highly involved in managing their child's disease on a daily basis, especially parents of affected children who are very young and more highly dependent upon parental caretaking.

It is not surprising that the experience of managing a child's diabetes can be demanding, overwhelming, and stressful for some parents, and may even significantly impair parental psychosocial well being. Further, difficulties achieving proper diabetes control have been reported to occur among parents of children of all ages, including parents of those who are very young.

Operationally, these psychosocial well being and diabetes outcomes can be examined by assessing: (1) parental symptoms of depression, anxiety, diabetes parenting stress, and perceived social support, and (2) metabolic control, which may be measured with the quarterly HbA1C counts.

As children diagnosed with Type 1 diabetes at a very young age may be at an increased risk for the development of long-term behavioral and medical complications due to the aforementioned difficulties (on the part of their parents), more research is needed to understand and treat the leading contributors to diabetes-related parental distress (depression, anxiety, stress, social support) and medical outcomes among this growing subgroup.

Recent findings indicate that responsibility for diabetes management falls heavily on mothers, who report performing 79% of their children's injections and 70% of blood glucose checks (Mednick, 2005). The majority of families do not receive outside child care assistance and report feeling overwhelmed. Parents report high levels of pediatric parenting stress difficulty, as well as moderate symptoms of anxiety. The current study aims to expand such preliminary findings and specifically examine the effects of a newly-developed parenting support program for parents of young children with Type 1 diabetes. The utility of the intervention will be evaluated. It is hypothesized that parents completing the parent support program will report lower levels of psychosocial distress and improved quality of life. It is hypothesized that the children of participating parents will also demonstrate improved quality of life and metabolic control.

Evaluating this intervention is a first step in the long-term goal of improving diabetes health outcomes for young children. Understanding the usefulness of this intervention can help us to further refine intervention programs for parents of young children with Type 1 diabetes that best meet their unique needs and risks.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 6 months prior to enrollment
* Seen for diabetes care at Children's National or Virginia Commonwealth
* Child ages 1-6

Exclusion Criteria:

* Non-English speaking primary caregiver
* Child with significant developmental delay

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Glycemic variability | baseline, 1, 6, and 12 months post intervention

SECONDARY OUTCOMES:
Parent Quality of Life | baseline, 1, 6, and 12 months post intervention
Child Quality of Life | baseline, 1, 6, and 12 months post intervention
Hemoglobin A1C | 6 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Randi Streisand, Ph.D., Principal Investigator — Children's National Research Institute
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Virginia Commonwealth University, Richmond, Virginia